CLINICAL TRIAL: NCT03444376
Title: A Multi-Center, Open-label Phase Ib-II Trial of the Combination of GX-188E Vaccination and Pembrolizumab in Patients With Advanced, Non-Resectable HPV Type 16 and/or 18 Positive Cervical Cancer
Brief Title: The Combination of GX-188E Vaccination and Pembrolizumab in Patients With HPV 16 and/or 18+ Advanced Cervical Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Genexine, Inc. (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GX-188E-005; MK-3475-567 (Other: Merck Sharp & Dohme LLC); KEYNOTE-567 (Other: Merck Sharp & Dohme LLC)
Record Dates: First submitted 2018-01-25; First posted 2018-02-23 (Actual); Results first posted 2025-07-30 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Cervical Cancer
Keywords: KEYTRUDA®; pembrolizumab; GX-188E; TDS-IM device; KEYNOTE-567
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — GX-188 vaccine; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- GX-188E, KEYTRUDA® (Experimental): GX-188E: 1st day of week 1,2,4,7,13,19, 46/ 2mg KEYTRUDA® : Day 1 q3 weeks/ 200mg
  Interventions: Drug: GX-188E; Drug: KEYTRUDA®

INTERVENTIONS:
Drug: GX-188E — GX-188E (1.0mg/0.5ml/vial), Intramuscular administration using electroporator, Ichor TDS-IM device
  Other Names: tirvalimogene teraplasmid
Drug: KEYTRUDA® — pembrolizumab(100mg/4mL/vial), Intravenous administration
  Other Names: pembrolizumab

SUMMARY:
A Multi-Center, Open-label Phase Ib-II Trial of the Combination of GX-188E Vaccination and Pembrolizumab in Patients with Advanced, Non-Resectable HPV-Positive Cervical Cancer

DETAILED DESCRIPTION:
This is an open-label Phase Ib-II trial to evaluate the safety and efficacy of GX-188E (IM administration using Ichor TDS-IM device) + pembrolizumab (P) in patients with advanced HPV-16+ or HPV-18+ cervical cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must be female and age ≥ 18 years (19 years for Korean sites)
2. Patients with histologically confirmed advanced or metastatic HPV-positive (HPV-16 or HPV-18) cervical cancer, who have disease progression after treatment with all available therapies for metastatic disease that are known to confer clinical benefit, or are intolerant to treatment, or refuse standard treatment.
3. Eastern Cooperative Oncology Group (ECOG) Performance Status of 0-1
4. Life Expectancy of at least 6 months
5. Patients must agree to provide either an archival tumor tissue sample or fresh biopsy sample for baseline biomarker tissue analyses, including staining for PD-L1. If archival tissue is not available and the patient does not have biopsy-accessible tumor lesions, the patient will be excluded.

Exclusion Criteria:

1. Patient has disease that is suitable for local therapy administered with curative intent.
2. Patient has a known additional malignancy that is progressing or has required active treatment within the past 3 years.
3. Patient is expected to require any other form of antineoplastic therapy while on study; including systemic chemotherapy, radiation therapy (except for palliative purposes) biological therapy, or immunotherapy not specified in this protocol.
4. Patient has a history of active central nervous system (CNS) metastases and/or carcinomatous meningitis.
5. Patients have received prior therapy with an anti-PD-1, anti-PD-L1, or anti PD-L2 agent or with an agent directed to another stimulatory or co-inhibitory T-cell receptor (e.g., CTLA-4, OX 40, CD137) and was discontinued from that treatment due to a Grade 3 or higher immune-related Adverse Event (irAE)
6. Patients with active autoimmune disease requiring systemic immunosuppressive treatment within the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (eg, thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment and is allowed.
7. Patients has had an allogeneic solid organ or allogeneic bone marrow transplant

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2018-06-19 (Actual); Primary Completion 2022-04-29 (Actual); Study Completion 2023-12-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Soo-Young Hur, M.D, Principal Investigator — The Catholic University of Korea
Locations (9):
- South Korea (9):
  - Inje University Busan Paik Hospital, Busan
  - Keimyung University Dongsan Medical Center, Daegu
  - National Cancer Center, Gyeonggi-do
  - Seoul National University Bundang Hospital, Gyeonggi-do
  - Severance Hospital, Yonsei University Health System, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - The Catholic University of Korea Seoul St. Mary's Hospital, Seoul
  - Korea University Guro Hospital, Seoul

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lim MC, Choi YJ, Hur SY, Kim YM, No JH, Kim BG, Cho CH, Kim SH, Jeong DH, Lee JK, Kim JH, Choi YJ, Woo JW, Sung YC, Park JS. GX-188E DNA vaccine plus pembrolizumab in HPV 16- and/or 18-positive recurrent or advance cervical cancer: a phase 2 trial. EClinicalMedicine. 2024 Jul 13;74:102716. doi: 10.1016/j.eclinm.2024.102716. eCollection 2024 Aug. PMID 39823099
- [Derived] Youn JW, Hur SY, Woo JW, Kim YM, Lim MC, Park SY, Seo SS, No JH, Kim BG, Lee JK, Shin SJ, Kim K, Chaney MF, Choi YJ, Suh YS, Park JS, Sung YC. Pembrolizumab plus GX-188E therapeutic DNA vaccine in patients with HPV-16-positive or HPV-18-positive advanced cervical cancer: interim results of a single-arm, phase 2 trial. Lancet Oncol. 2020 Dec;21(12):1653-1660. doi: 10.1016/S1470-2045(20)30486-1. PMID 33271094

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 90 subjects were enrolled, of which 25 subjects were considered as screen failures.
  Of 90 Screened, 65 met Inclusion/Exclusion Criteria and were Randomized to treatment.
Pre-assignment Details: Subjects were enrolled in three Parts; 6 subjects in Part A, 31 subjects in Part B (6 rolled over from Part A to Part B) and 65 subjects in Part C (6 rolled over from Part A and 25 from Part B) were enrolled.
  Of the 25 subjects enrolled during Part B period, 1 subject completed Part B and rolled over to Part C to continue the study, but died during Part C period. Therefore, this subject was counted as 'Completed' for Part B period, but 'Not Completed due to Death' for Part C period.
Groups:
- Single Arm (GX-188E + Pembrolizumab): Assigned Participants: 65 subjects
  Intervention: Receiving GX-188E at 2 mg (1mg/site x 2 vaccination sites) at week 1, 2, 4, 7, 13, 19, 46 and 200 mg Pembrolizumab on Day 1 q3 weeks.
  Design: In Part A, the first 6 subjects were enrolled and evaluated for the first 3 weeks for DLTs. No additional subjects were enrolled until all subjects in Part A completed the DLT window and the treatment regimen was deemed safe. If none or only 1 of the first 6 subjects experienced a DLT the study was moved into Part B.
  Part B employed a Simon Two-Stage design to evaluate the anti-tumor efficacy of the GX-188E + pembrolizumab at the recommended Phase 2 schedule established as tolerable in Part A. In Stage 1 of Part B, 15 subjects were treated. These might have included any subjects from Part A, who did not experience a DLT, received the recommended Phase 2 treatment regimen, and who were considered evaluable for efficacy. If at least 3 efficacy evaluable subjects from Part B Stage 1 had objective responses within the first 24 weeks of treatment, an additional 13 subjects were enrolled, for a total of 28 efficacy evaluable subjects.
  For Part C, if at least 8 of the 28 subjects enrolled in Part B, experienced an objective response who were considered evaluable for efficacy, it was considered that ORR satisfied the criteria for study expansion and additional subjects were enrolled in Part C to evaluate the efficacy further in larger population.
Period: Part A
Arm/Group | Single Arm (GX-188E + Pembrolizumab)
Started | 6
Completed | 2
Not Completed | 4
Not completed — Disease relapse or Progression | 1
Not completed — Withdrawal by Subject | 2
Not completed — Adverse Event | 1
Period: Part B
Arm/Group | Single Arm (GX-188E + Pembrolizumab)
Started | 31
Completed | 8
Not Completed | 23
Not completed — Disease relapse or Progression | 18
Not completed — Withdrawal by Subject | 2
Not completed — Adverse Event | 2
Not completed — Physician Decision | 1
Period: Part C
Arm/Group | Single Arm (GX-188E + Pembrolizumab)
Started | 65
Completed | 12
Not Completed | 53
Not completed — Disease relapse or Progression | 43
Not completed — Withdrawal by Subject | 5
Not completed — Adverse Event | 2
Not completed — Physician Decision | 2
Not completed — Death | 1

BASELINE CHARACTERISTICS:
Arm/Group | GX-188E, KEYTRUDA®
Number analyzed (Participants) | 65
Age, Categorical [Count of Participants; unit: Participants] — Population: Six subjects in Part A, 31 subjects in Part B (6 subjects rolled over from Part A to Part B) and 65 subjects in Part C (6 subjects rolled over from Part A and 25 subjects from Part B) were enrolled
  Participants
    Part A: number analyzed (Participants) | 6
    Part A: <=18 years | 0
    Part A: Between 18 and 65 years | 5
    Part A: >=65 years | 1
    Part B: number analyzed (Participants) | 31
    Part B: <=18 years | 0
    Part B: Between 18 and 65 years | 29
    Part B: >=65 years | 2
    Part C: <=18 years | 0
    Part C: Between 18 and 65 years | 59
    Part C: >=65 years | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 65
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 65
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
PD-L1 expression status [Count of Participants; unit: Participants] — Population: Six subjects in Part A, 31 subjects in Part B (6 subjects rolled over from Part A to Part B) and 65 subjects in Part C (6 subjects rolled over from Part A and 25 subjects from Part B) were enrolled.
  Participants
    Part A: number analyzed (Participants) | 6
    Part A: Positive (≥1 CPS) | 0
    Part A: Negative (<1 CPS) | 6
    Part B: number analyzed (Participants) | 31
    Part B: Positive (≥1 CPS) | 15
    Part B: Negative (<1 CPS) | 16
    Part C: Positive (≥1 CPS) | 39
    Part C: Negative (<1 CPS) | 26
Histologic Type [Count of Participants; unit: Participants] — Population: Six subjects in Part A, 31 subjects in Part B (6 subjects rolled over from Part A to Part B) and 65 subjects in Part C (6 subjects rolled over from Part A and 25 subjects from Part B) were enrolled.
  Participants
    Part A: number analyzed (Participants) | 6
    Part A: Squamous Cell Carcinoma | 3
    Part A: Adenocarcinoma | 3
    Part B: number analyzed (Participants) | 31
    Part B: Squamous Cell Carcinoma | 23
    Part B: Adenocarcinoma | 8
    Part C: Squamous Cell Carcinoma | 50
    Part C: Adenocarcinoma | 15
HPV type [Count of Participants; unit: Participants] — Population: Six subjects in Part A, 31 subjects in Part B (6 subjects rolled over from Part A to Part B) and 65 subjects in Part C (6 subjects rolled over from Part A and 25 subjects from Part B) were enrolled.
  Participants
    Part A: number analyzed (Participants) | 6
    Part A: HPV-16 | 3
    Part A: HPV-18 or both | 3
    Part B: number analyzed (Participants) | 31
    Part B: HPV-16 | 24
    Part B: HPV-18 or both | 7
    Part C: HPV-16 | 49
    Part C: HPV-18 or both | 16

OUTCOME MEASURES:

1. Primary Outcome: DLT Evaluation for Safety and Tolerability(Part A)
Description: Patient will be evaluated for the first 21 days for dose-limiting toxicities.
Time Frame: within 21days
Population: The first 6 subjects (Part A) were enrolled and evaluated for the first 3 weeks (prior to Week 4 Day 1 visit) for DLTs. No additional subjects were enrolled until all subjects in Part A completed the DLT window and the investigational treatment regimen was deemed safe.
Measure: Number; unit: participants
Arm/Group | GX-188E, KEYTRUDA®
Number analyzed (Participants) | 6
participants | 0

2. Primary Outcome: ORR for Efficacy (Part B&C)
Description: ORR within 24 weeks (ORR24) evaluated by RECIST v1.1
Time Frame: within 24 weeks
Population: All efficacy analyses included 60 subjects from the Efficacy Evaluable Population. Safety analyses included 65 subjects. Five subjects were excluded from efficacy analysis for receiving less than 45 days of treatment without experiencing any DLT. The efficacy population comprised 6 subjects in Part A, 29 in Part B (including 6 from Part A), and 60 in Part C (including 6 from Part A and 23 from Part B).
Measure: Number (95% Confidence Interval); unit: percentage of responders
Arm/Group | GX-188E, KEYTRUDA®
Number analyzed (Participants) | 60
percentage of responders
  Part B: number analyzed (Participants) | 29
  Part B | 41.4 [25.89 to 100.00]
  Part C | 35.0 [22.93 to 47.07]

3. Secondary Outcome: ORR for Efficacy (Part A)
Description: Overall Response Rate within 24 weeks (ORR24) by RECIST v1.1 and immune-related Response Criteria (irRC)
Time Frame: within 24 weeks
Population: All efficacy analyses were carried out using the 60 in the Efficacy Evaluable Population, respectively, and ORR24 analysis was performed for 6 subjects in the Part A group.
Measure: Number (95% Confidence Interval); unit: percentage of responders
Arm/Group | GX-188E, KEYTRUDA®
Number analyzed (Participants) | 6
percentage of responders | 50.0 [11.81 to 88.19]

4. Secondary Outcome: BORR (Part B&C)
Description: Best Overall Response Rate(BORR) by RECIST v1.1
Time Frame: up to 1 year
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of responders
Arm/Group | GX-188E, KEYTRUDA®
Number analyzed (Participants) | 60
percentage of responders
  Part A: number analyzed (Participants) | 6
  Part A | 50.0 [11.81 to 88.19]
  Part B: number analyzed (Participants) | 29
  Part B | 41.4 [23.52 to 61.06]
  Part C | 35.0 [22.93 to 47.07]

5. Secondary Outcome: Time-to-Best Response
Description: Time-to-Best Response by RECIST v1.1 and iRECIST
Time Frame: up to 1 year
Population: as for outcome 2
Measure: Median (90% Confidence Interval); unit: Months
Arm/Group | GX-188E, KEYTRUDA®
Number analyzed (Participants) | 60
Months
  Part A: number analyzed (Participants) | 6
  Part A | 2.07 [2.07 to NA] — Upper limit of 95% CI could not be calculated due to low number of participants with events.
  Part B: number analyzed (Participants) | 29
  Part B | 2.10 [2.04 to 4.01]
  Part C | 2.10 [2.07 to 3.02]

6. Secondary Outcome: Duration of Response (DOR)
Description: Duration of Response (DOR) by RECIST v1.1 and iRECIST
Time Frame: up to 1 year
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | GX-188E, KEYTRUDA®
Number analyzed (Participants) | 60
Months
  Part A: number analyzed (Participants) | 6
  Part A | NA [2.40 to NA] — Median and Upper limit of 95% CI could not be calculated due to low number of participants with events.
  Part B: number analyzed (Participants) | 29
  Part B | 5.78 [2.40 to NA] — Upper limit of 95% CI could not be calculated due to low number of participants with events.
  Part C | NA [5.32 to NA] — Median and Upper limit of 95% CI could not be calculated due to low number of participants with events.

7. Secondary Outcome: Progression-Free Survival (PFS)
Description: 6month- PFS by RECIST v1.1 and iRECIST
Time Frame: up to 6 months
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | GX-188E, KEYTRUDA®
Number analyzed (Participants) | 60
Months
  Part A: number analyzed (Participants) | 6
  Part A | 4.25 [2.04 to NA] — Upper limit of 95% CI could not be calculated due to low number of participants with events.
  Part B: number analyzed (Participants) | 29
  Part B | 4.14 [2.07 to 8.38]
  Part C | 4.40 [2.14 to 8.31]

8. Secondary Outcome: Overall Survival (OS)
Description: Overall Survival (OS) by RECIST v1.1 and iRECIST
Time Frame: up to 1 year
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | GX-188E, KEYTRUDA®
Number analyzed (Participants) | 60
Months
  Part A: number analyzed (Participants) | 6
  Part A | 15.54 [3.48 to NA] — Due to low number of events, the upper limit of 95% CI from Kaplan-Meier survival curves could not derived.
  Part B: number analyzed (Participants) | 29
  Part B | 14.42 [8.97 to NA] — Due to low number of events, the upper limit of 95% CI from Kaplan-Meier survival curves could not derived.
  Part C | 23.79 [14.03 to NA] — Due to low number of events, the upper limit of 95% CI from Kaplan-Meier survival curves could not derived.

ADVERSE EVENTS:
Time Frame: 24 months
Arm/Group | GX-188E, KEYTRUDA®
All-Cause Mortality (participants affected / at risk) | 31/65
Serious Adverse Events (participants affected / at risk) | 25/65
Other Adverse Events (participants affected / at risk) | 54/65
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | GX-188E, KEYTRUDA® (N=65)
Urinary tract infection (Infections and infestations) | 7
Pneumonia (Infections and infestations) | 2
Appendicitis (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 1
Kidney infection (Infections and infestations) | 1
Lymphangitis (Infections and infestations) | 1
Ophthalmic herpes zoster (Infections and infestations) | 1
Peritonitis (Investigations) | 1
Pyrexia (General disorders) | 3
Asthenia (General disorders) | 2
Acute kidney injury (Renal and urinary disorders) | 1
Azotaemia (Renal and urinary disorders) | 1
Hydronephrosis (Renal and urinary disorders) | 1
Urinary tract obstruction (Renal and urinary disorders) | 1
Urogenital fistula (Renal and urinary disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Colitis ischaemic (Gastrointestinal disorders) | 1
Haematochezia (Gastrointestinal disorders) | 1
Mechanical ileus (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Pericardial effusion (Cardiac disorders) | 1
Blood creatinine increased (Investigations) | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1
Small intestine carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Vaginal fistula (Reproductive system and breast disorders) | 1
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | GX-188E, KEYTRUDA® (N=65)
Abdominal pain (Gastrointestinal disorders) | 6
Constipation (Gastrointestinal disorders) | 7
Diarrhoea (Gastrointestinal disorders) | 7
Nausea (Gastrointestinal disorders) | 6
Vomiting (Gastrointestinal disorders) | 6
Dyspepsia (Gastrointestinal disorders) | 3
Abdominal distension (Gastrointestinal disorders) | 2
Chronic gastritis (Gastrointestinal disorders) | 2
Urinary tract infection (Infections and infestations) | 6
Herpes zoster (Infections and infestations) | 4
Pneumonia (Infections and infestations) | 3
Conjunctivitis (Infections and infestations) | 2
Cystitis (Infections and infestations) | 3
Nasopharyngitis (Infections and infestations) | 2
Blood creatinine increased (Investigations) | 8
Alanine aminotransferase increased (Investigations) | 5
Aspartate aminotransferase increased 0 (Investigations) | 5
Neutrophil count decreased (Investigations) | 3
Blood thyroid stimulating hormone increased (Investigations) | 2
Weight decreased (Investigations) | 2
Pyrexia (General disorders) | 8
Asthenia (General disorders) | 5
Fatigue (General disorders) | 3
Oedema peripheral (General disorders) | 3
Hypoalbuminaemia (Metabolism and nutrition disorders) | 6
Decreased appetite (Metabolism and nutrition disorders) | 4
Hypomagnesaemia (Metabolism and nutrition disorders) | 4
Hypoglycaemia (Metabolism and nutrition disorders) | 2
Hypokalaemia (Metabolism and nutrition disorders) | 2
Hypocalcaemia (Metabolism and nutrition disorders) | 2
Anaemia (Blood and lymphatic system disorders) | 19
Cough (Respiratory, thoracic and mediastinal disorders) | 8
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 3
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2
Productive cough (Respiratory, thoracic and mediastinal disorders) | 2
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 4
Back pain (Musculoskeletal and connective tissue disorders) | 2
Neck pain (Musculoskeletal and connective tissue disorders) | 3
Flank pain (Musculoskeletal and connective tissue disorders) | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2
Dizziness (Nervous system disorders) | 4
Headache (Nervous system disorders) | 5
Rash (Skin and subcutaneous tissue disorders) | 5
Pruritus (Skin and subcutaneous tissue disorders) | 4
Urticaria (Skin and subcutaneous tissue disorders) | 3
Dermatitis (Skin and subcutaneous tissue disorders) | 3
Hypothyroidism (Endocrine disorders) | 10
Thyroiditis (Endocrine disorders) | 3
Acute kidney injury (Renal and urinary disorders) | 2
Hydronephrosis (Renal and urinary disorders) | 2
Haematuria (Renal and urinary disorders) | 3
Dry eye (Eye disorders) | 3
Lymphoedema (Vascular disorders) | 5
Hypertension (Vascular disorders) | 2
Pelvic pain (Reproductive system and breast disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2022-08-29): https://cdn.clinicaltrials.gov/large-docs/76/NCT03444376/Prot_000.pdf
  • Statistical Analysis Plan (2022-09-05): https://cdn.clinicaltrials.gov/large-docs/76/NCT03444376/SAP_001.pdf